CLINICAL TRIAL: NCT06011863
Title: Effectiveness Comparison Of Preemptive Single-Dose Thoracic Epidural Analgesia And Erector Spinae Plane Block For Thoracotomy Analgesia In Thoracic Surgery
Brief Title: Comparison of Pain Relief Efficacy of Epidural Analgesia and Erector Spinae Plane Block Before Thoracotomy Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Saglik Bilimleri Universitesi Gazi Yasargil Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Fatma Acil, Principal Investigator, Saglik Bilimleri Universitesi Gazi Yasargil Training and Research Hospital
Other Study IDs: 10.21.2022/216
Record Dates: First submitted 2023-08-08; First posted 2023-08-25 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-10

CONDITIONS: Thoracotomy Surgery
MeSH Terms: interventions — Tea

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group TEA (Thoracic Epidural Analgesia): Group TEA (Thoracic Epidural Analgesia): Thoracic Epidural Application: The epidural area will be accessed from the 7th (T7)-8th (T8) level of the thoracic vertebral midline with an 18 gauge (G) epidural needle using the hanging drip technique. After 2 ml of 2% lidocaine is administered and no spinal effect is observed, a mixture of morphine and local anaesthetic 3-4 mg morphine hydrochloride + 5 ml 0.5% bupivacaine + 2 ml 0.9% saline will be administered through the epidural needle at once and the epidural needle will be withdrawn and sterile dressing will be applied.
  Interventions: Procedure: Thoracic Epidural Analgesia
- Grup ESP ( Erector spinae plane block): Group ESP: Before induction of anaesthesia, the patient is placed on the operating table and placed in a forward tilted position. Asepsis and antisepsis conditions are provided. The linear USG probe is moved approximately 2-3 cm lateral to the spinous process T5 - T6 level on the side to be operated. The trapezius, rhomboid major and erector spinae muscles will be identified to find the correct probe position. A 22 gauge , 50 mm or 22 gauge 80 mm single shot nerve blocks needle will be inserted through the skin in a cranio-caudal direction. With the needle resting on the transverse process, the plane between the erector spinae muscle and the transverse process will be verified by hydrodissection with 5 ml saline solution. Then 20 ml of 0.25% bupivacaine will be injected. The ESP block will be considered successful if the local anaesthetic spreads linearly up to the T8 - T9 level. The patient will then be placed in the supine position and general anaesthesia will be administered.
  Interventions: Procedure: Erector spinae plane block

INTERVENTIONS:
Procedure: Thoracic Epidural Analgesia — Thoracic Epidural Application: The epidural area will be accessed from the 7th (T7)-8th (T8) level of the thoracic vertebral midline with an 18 gauge (G) epidural needle using the hanging drip technique. After 2 ml of 2% lidocaine is administered and no spinal effect is observed, a mixture of morphine and local anaesthetic 3-4 mg morphine hydrochloride + 5 ml 0.5% bupivacaine + 2 ml 0.9% saline will be administered through the epidural needle at once and the epidural needle will be withdrawn and sterile dressing will be applied.
  Groups: Group TEA (Thoracic Epidural Analgesia)
Procedure: Erector spinae plane block — Before induction of anaesthesia, the patient is placed on the operating table and placed in a forward tilted position. Asepsis and antisepsis conditions are provided. The linear USG probe is moved approximately 2-3 cm lateral to the spinous process T5 - T6 level on the side to be operated. The trapezius, rhomboid major and erector spinae muscles will be identified to find the correct probe position. A 22 gauge 50 mm or 22 gauge 80 mm single shot nerve blocks needle will be inserted through the skin in a cranio-caudal direction. With the needle resting on the transverse process, the plane between the erector spinae muscle and the transverse process will be verified by hydrodissection with 5 ml saline solution. Then 20 ml of 0.25% bupivacaine will be injected. The ESP block will be considered successful if the local anaesthetic spreads linearly up to the T8 - T9 level. The patient will then be placed in the supine position and general anaesthesia will be administered.
  Groups: Grup ESP ( Erector spinae plane block)

SUMMARY:
In patients who will undergo open thoracic surgery, two different types of drugs will be administered to volunteer patients before surgery in order to relieve postoperative pain, facilitate breathing and reduce hospitalization time. The pain intensity, respiratory capacity, the amount of opioid analgesic needed during and after surgery, side effects such as nausea-vomiting, low blood pressure and shortness of breath will be evaluated.

DETAILED DESCRIPTION:
Group Thoracic Epidural Analgesia (TEA): Thoracic Epidural Application: The epidural area will be accessed from the 7th (T7)-8th (T8) level of the thoracic vertebral midline with an 18 gauge (G) epidural needle using the hanging drip technique. After 2 ml of 2% lidocaine is administered and no spinal effect is observed, a mixture of morphine and local anaesthetic 3-4 mg morphine hydrochloride + 5 ml 0.5% bupivacaine + 2 ml 0.9% saline will be administered through the epidural needle at once and the epidural needle will be withdrawn and sterile dressing will be applied.

* The mode of presentation will be face-to-face and individually.
* The intervention will be performed by an anaesthetist with at least 5 years of experience.
* The stages of the intervention will be verbally explained in detail to participants prior to the intervention.
* The patient will be taken to the operating table and electrocardiographic, oxygen saturation with pulse oximetry and non-invasive blood pressure monitoring with automatic manometer will be performed.

The intervention will be administered only once, 3-4 mg of morphine hydrochloride + 5 ml of 0.5 % bupivacaine + 2 ml of 0.9 % saline into the epidural space.

* Immediately before induction of anaesthesia, the patient will be seated and after appropriate sterilisation conditions are provided, the thoracic epidural space will be reached and the analgesic mixture will be given once and the space will be exited.
* Immediately after sterile dressing of the intervention site, the patient will be placed supine and standard general anaesthesia will be applied.
* The intervention will be performed in the thoracic surgery room of our hospital operating theatre.

Grup Erector spinae plane block (ESP): Before induction of anaesthesia, the patient will be placed on the operating table and placed in a forward tilted position. Asepsis and antisepsis conditions will be fulfilled.

The linear ultrasonogram (USG) probe will first be placed in the sagittal plane to visualise the vertebral spinous process. Then the linear probe was moved approximately 2-3 cm lateral to the spinous process T5 - T6 level on the side to be operated on, and the probe will be rotated 90 degrees to the longitudinal plane to visualise the transverse process. The trapezius, rhomboid major and erector spinae muscles will be identified to find the correct probe position. A 22 gauge, 50 mm or 22 gauge 80 mm single shot nerve blocks needle will be inserted through the skin in a cranio-caudal direction. With the needle resting on the transverse process, the plane between the erector spinae muscle and the transverse process will be verified by hydrodissection with 5 ml saline solution. Then, 20 ml of 0.25% bupivacaine will be injected. The ESP block will be considered successful if the local anaesthetic spreads linearly up to the T8 - T9 level. The patient will then be placed in the supine position and general anaesthesia will be administered.

* The mode of presentation will be face-to-face and individually.
* The intervention will be performed by an anaesthetist with at least 5 years of experience.
* The stages of the intervention will be verbally explained in detail to participants prior to the intervention.
* The patient will be taken to the operating table and electrocardiographic, oxygen saturation with pulse oximetry and non-invasive blood pressure monitoring with automatic manometer will be performed.
* The intervention will be performed only once on the side of the surgical incision and 20 ml of 0.25% bupivacaine will be injected once into the relevant area.
* Immediately before induction of anaesthesia, the patient will be seated and after appropriate sterilisation conditions are provided, the fascia of the erector spina muscle will be reached under ultrasound guidance and the analgesic solution will be given to this area only once and the cavity will be exited.
* Immediately after sterile dressing of the intervention site, the patient will be placed supine and standard general anaesthesia will be applied.
* The intervention will be performed in the thoracic surgery room of our hospital operating theatre.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) I-III physical condition
* who were to undergo thoracotomy

Exclusion Criteria:

* patients with acute infection,
* coagulation disorder,
* morbid obesity (Body Mass Index (BMI) > 35),
* drug allergy
* history of chronic pain,
* long-term opioid use,
* history of psychiatric illness,
* emergency surgeries

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients undergoing thoracotomy surgery
Sampling Method: Probability Sample
Enrollment: 42 (Estimated)
Dates: Start 2023-10-03 (Actual); Primary Completion 2023-12-27 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) | At the minute of admission to the postoperative care unit (PACU), in the first 30 minutes after surgery, in the 2nd hour after surgery, in the 6th hour after surgery, in the 12th hour after surgery, at the 24th hour after surgery
  The visual analog scale (VAS) is a validated, subjective measure for acute and chronic pain. Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between "no pain" and "worst pain."

SECONDARY OUTCOMES:
Inspiratory spirometry test | At the minute of admission to the postoperative care unit (PACU),in the first 30 minutes after surgery, in the 2nd hour after surgery, in the 6th hour after surgery, in the 12th hour after surgery, at the 24th hour after surgery
  The inspiratory spirometry test will be performed and the inspiratory flow rate calculated according to the number of rising balls will be recorded (1 ball = 600 ml, 2 balls = 900 ml, 3 balls = 1200 ml).
Postoperative nausea and/or vomiting (PONV) | At the minute of admission to the postoperative care unit (PACU), in the first 30 minutes after surgery, in the 2nd hour after surgery, in the 6th hour after surgery, in the 12th hour after surgery, at the 24th hour after surgery
  Questioning about the presence/absence of nausea and/or vomiting in the postoperative period
Amount of fentanyl used intraoperatively | during surgery
  Amount of fentanyl used intraoperatively (µg)
Amount of tramadol used postoperatively | during the postoperative 24 hour
  Amount of tramadol used postoperatively (milligrams)
Surgery duration | at the end of surgery
  Time in hours from the start of the surgical incision until the last surgical suture is placed
Anesthesia duration | as soon as the patient is extubated
  time in hours from induction of anaesthesia to extubation
Length of stay in intensive care | It is assessed for up to 12 months from the date of surgery to the date of the first documented progression or the date of death from any cause, whichever comes first
  Length of stay in intensive care unit in days
Length of hospital stay | It is assessed for up to 12 months from the date of surgery to the date of the first documented progression or the date of death from any cause, whichever comes first
  days of hospitalisation after the operation

CONTACTS AND LOCATIONS:
Overall Officials: Fatma Acil, Principal Investigator — Saglik Bilimleri Universitesi Gazi Yasargil Training and Research Hospital
Locations (1):
- Saglik Bilimleri Universitesi Gazi Yasargil Training and Research Hospital, Diyarbakır, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Zhang Y, Fu Z, Fang T, Wang K, Liu Z, Li H, Jiang W, Cao X. A comparison of the analgesic efficacy of serratus anterior plane block vs. paravertebral nerve block for video-assisted thoracic surgery: a randomized controlled trial. Wideochir Inne Tech Maloinwazyjne. 2022 Mar;17(1):134-142. doi: 10.5114/wiitm.2021.105725. Epub 2021 Apr 30. PMID 35251398